CLINICAL TRIAL: NCT01727258
Title: Evaluation of an Experimental Mouth Rinse Device for Relieving Dentinal Hypersensitivity
Brief Title: A Test on a New Experimental Mouth Rinse for Relieving Tooth Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: KOXDHY0008
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-04

CONDITIONS: Dentin Sensitivity
Keywords: Tooth Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mouth Rinse (Experimental): Twice daily for 28 days, brush in usual manner for at least one minute using at least a one-inch strip of Fluoride Toothpaste provided. Rinse with water after brushing teeth. Then rinse for 60 seconds with 10 mL of the experimental Mouth Rinse 12027-033 (KOX).
  Interventions: Device: Mouth Rinse; Drug: Fluoride Toothpaste
- Fluoride Toothpaste (Active Comparator): Twice daily for 28 days, brush in usual manner for at least one minute using at least a one-inch strip of the Fluoride Toothpaste (NEG) provided.
  Interventions: Drug: Fluoride Toothpaste
- Potassium Nitrate Toothpaste (Active Comparator): Twice daily for 28 days, brush in usual manner for at least one minute using at least a one-inch strip of the Potassium Nitrate Toothpaste (POS) provided.
  Interventions: Drug: Potassium Nitrate Toothpaste

INTERVENTIONS:
Device: Mouth Rinse — Mouth rinse 12027-033 used twice daily for 28 days after brushing.
  Arms: Mouth Rinse
Drug: Fluoride Toothpaste — Fluoride Toothpaste used daily for 28 days.
  Other Names: Colgate® Cavity Protection Regular
  Arms: Fluoride Toothpaste; Mouth Rinse
Drug: Potassium Nitrate Toothpaste — Potassium Nitrate Toothpaste used daily for 28 days.
  Other Names: Sensodyne® Original
  Arms: Potassium Nitrate Toothpaste

SUMMARY:
This study is for people with sensitive teeth and involves going to the dentist for 4 visits over 6 weeks. At each visit the dentist will look at the mouth, teeth, tongue and gums of subjects, and check for sensitive teeth.

During the first 2 weeks, participants will brush their teeth two times a day with the fluoride toothpaste provided.

Then, if they qualify to continue in the study, participants will be assigned to a treatment group. All the groups will get toothpaste currently sold on the market, and one group will get a mouthwash with an experimental ingredient to use as well. Subjects will have an equal chance of being assigned to any one of the three groups.

For the next 4 weeks, subjects will use their assigned products according to the directions provided. At Visit 1 subjects will be supervised while they brush their teeth to ensure they understand the directions. They will also have supervised use of the product at Visit 2.

We will see if the mouthwash helps to reduce tooth sensitivity during the study.

DETAILED DESCRIPTION:
This study will consist of run-in and treatment phases. To qualify for the study, subjects must meet the inclusion/exclusion criteria and return tactile sensitivity scores within protocol-specified parameters at both the screening and baseline visits.

Run-in will consist of a 2-week period during which subjects will use a sodium fluoride dentifrice. At the start of the first phase, subjects will attend a Screening Visit. They will participate in the informed consent process, complete a medical/dental history, and be evaluated for tactile sensitivity to Yeaple probe and response to a cold air stimulus.

Subjects who qualify through screening will begin a run-in period that will last approximately two weeks. The run-in period will be followed by a Baseline visit. Subjects who continue to qualify through Baseline will be randomized to one of three treatment groups.

During the four-week treatment period, all subjects will brush their teeth twice daily for at least one minute in their usual manner, with their assigned toothpaste. After brushing, subjects assigned to the mouth rinse group will rinse with water, and then rinse with 10 mL of the experimental mouth rinse for 60 seconds.

The study duration is approximately six weeks with each subject visiting the clinical site six times.

Adverse events will be observed and collected by querying each subject at each visit for new or continuing symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Good general and oral health without any known allergy to commercial dental products or cosmetics
* Evidence of a personally signed and dated informed consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial
* Willingness to use the assigned products according to instructions, availability for appointments, and likelihood of completing the clinical trial
* Dental condition appropriate for inclusion in the trial according to protocol-specified parameters and the professional opinion of the investigator
* Adequate oral hygiene (i.e. brush teeth daily and exhibit no signs of oral neglect

Exclusion Criteria:

* Medical condition or history, or use of drugs or treatments that could possibly compromise the safety of the research subject or the interpretation of results, per protocol or in the opinion of the investigator
* Use of home-care bleaching, whitening products or professional bleaching treatment within a protocol-specified time period
* Use of desensitizing agents within a protocol-specified time period
* Participation in a dental clinical trial involving oral care products within a protocol-specified time period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lynch, DMD, PhD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (1):
- BioSci Research America, Inc., Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Colgate Regular: Standard Sodium Fluoride Dentifrice (Negative Control) (UPC #035000513007).
- Sensodyne Toothpaste: 5% Potassium Nitrate Dentifrice (Positive Control) (UPC #310158077046).
- Potassium Oxalate Mouthrinse: Potassium Oxalate Mouthrinse (experimental group)(12027-033).
Period: Overall Study
Arm/Group | Colgate Regular | Sensodyne Toothpaste | Potassium Oxalate Mouthrinse
Started | 51 | 51 | 51
Completed | 49 | 48 | 50
Not Completed | 2 | 3 | 1
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Noncompliance with Study Drug | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colgate Regular | Sensodyne Toothpaste | Potassium Oxalate Mouthrinse | Total
Number analyzed (Participants) | 51 | 51 | 51 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (10.97) | 37.0 (11.56) | 39.9 (10.46) | 38.4 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 37 | 39 | 109
  Male | 18 | 14 | 12 | 44
Region of Enrollment [Number; unit: participants]
  USA | 51 | 51 | 51 | 153

OUTCOME MEASURES:

1. Primary Outcome: Mean Tactile Sensitivity Score at Week 4
Description: Tooth sensitivity was measured using a Yeaple probe. The force at which discomfort was felt by the participant was recorded on a scale of 10-80 grams. The score for each participant was calculated by averaging the scores for all study teeth for that participant.
Time Frame: 4 weeks
Population: Analysis was based on the Intent-to-Treat (ITT) analysis set, defined as all randomized participants who used at least one dose of the study product and had baseline and at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: grams of force
Arm/Group | Colgate Regular | Sensodyne Toothpaste | Potassium Oxalate Mouthrinse
Number analyzed (Participants) | 49 | 48 | 50
grams of force | 11.21 (1.221) | 23.81 (1.234) | 22.07 (1.210)
Statistical Analysis 1: Comparison: Colgate Regular vs Potassium Oxalate Mouthrinse; The null hypothesis was no difference in mean outcome between treatment groups. The alternative hypothesis was a difference in mean outcome between treatment groups; Test type: Superiority or Other; p < 0.001, ANCOVA — If Potassium Oxalate Mouthrinse is better than Colgate Regular (p<0.05), testing would proceed to comparison of Wk 2 Mean Tactile Sensitivity Scores between Potassium Oxalate Mouthrinse and Colgate Regular. Family-wise error was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = 10.85, 95% CI 2-sided [7.45 to 14.25], Standard Error of Mean 1.720
Statistical Analysis 2: Comparison: Sensodyne Toothpaste vs Potassium Oxalate Mouthrinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.314, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = -1.74, 95% CI 2-sided [-5.16 to 1.67], Standard Error of Mean 1.729
Statistical Analysis 3: Comparison: Colgate Regular vs Sensodyne Toothpaste; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = 12.60, 95% CI 2-sided [9.17 to 16.03], Standard Error of Mean 1.735

2. Primary Outcome: Mean Tactile Sensitivity Score at Week 2
Description: as for outcome 1
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: grams of force
Arm/Group | Colgate Regular | Sensodyne Toothpaste | Potassium Oxalate Mouthrinse
Number analyzed (Participants) | 50 | 49 | 50
grams of force | 11.09 (0.832) | 17.00 (0.840) | 17.18 (0.832)
Statistical Analysis 1: Comparison: Colgate Regular vs Potassium Oxalate Mouthrinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — If Potassium Oxalate Mouthrinse is better than Colgate Regular (p<0.05), testing would proceed to comparison of Wk 2 Mean Tactile Sensitivity Scores between Potassium Oxalate Mouthrinse and Sensodyne. Family-wise error was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = 6.08, 95% CI 2-sided [3.76 to 8.41], Standard Error of Mean 1.177
Statistical Analysis 2: Comparison: Sensodyne Toothpaste vs Potassium Oxalate Mouthrinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.881, ANCOVA — The significance threshold level was 0.05 (two-sided). Family-wise error was controlled at 0.05; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-2.16 to 2.52], Standard Error of Mean 1.183
Statistical Analysis 3: Comparison: Colgate Regular vs Sensodyne Toothpaste; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity (Yeaple probe) score; Mean Difference (Final Values) = 5.91, 95% CI 2-sided [3.57 to 8.24], Standard Error of Mean 1.182

3. Secondary Outcome: Mean Tactile Sensitivity VAS Score at Week 2
Description: Tooth sensitivity was measured using a Visual Analogue Scale (VAS). At each visit, participants rated their perception of the pain/discomfort experienced from the Yeaple probe by marking a single vertical line on a VAS scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm. The investigator recorded a VAS score of 0 mm for participants who did not experience discomfort at the maximum force of 80 grams. The score for each participant was calculated by averaging the scores for all study teeth for that participant.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Colgate Regular | Sensodyne Toothpaste | Potassium Oxalate Mouthrinse
Number analyzed (Participants) | 50 | 49 | 50
units on a scale (mm) | 43.80 (2.009) | 36.95 (2.020) | 37.08 (2.017)
Statistical Analysis 1: Comparison: Colgate Regular vs Potassium Oxalate Mouthrinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.020, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = -6.72, 95% CI 2-sided [-12.38 to -1.05], Standard Error of Mean 2.866
Statistical Analysis 2: Comparison: Sensodyne Toothpaste vs Potassium Oxalate Mouthrinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.964, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-5.52 to 5.78], Standard Error of Mean 2.860
Statistical Analysis 3: Comparison: Colgate Regular vs Sensodyne Toothpaste; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.017, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = -6.85, 95% CI 2-sided [-12.47 to -1.23], Standard Error of Mean 2.845

4. Secondary Outcome: Mean Tactile Sensitivity VAS Score at Week 4
Description: as for outcome 3
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Colgate Regular | Sensodyne Toothpaste | Potassium Oxalate Mouthrinse
Number analyzed (Participants) | 49 | 48 | 50
units on a scale (mm) | 38.38 (2.342) | 26.40 (2.353) | 31.45 (2.327)
Statistical Analysis 1: Comparison: Colgate Regular vs Potassium Oxalate Mouthrinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.039, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = -6.92, 95% CI 2-sided [-13.50 to -0.35], Standard Error of Mean 3.327
Statistical Analysis 2: Comparison: Sensodyne Toothpaste vs Potassium Oxalate Mouthrinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.130, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = 5.06, 95% CI 2-sided [-1.50 to 11.61], Standard Error of Mean 3.317
Statistical Analysis 3: Comparison: Colgate Regular vs Sensodyne Toothpaste; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean tactile sensitivity VAS score; Mean Difference (Final Values) = -11.98, 95% CI 2-sided [-18.53 to -5.43], Standard Error of Mean 3.313

5. Secondary Outcome: Mean Cold Air Stimulus VAS Score at Week 2
Description: Tooth sensitivity was measured using a Cold Air Stimulus. When being assessed, participants rated their perception of the pain/discomfort experienced when cold air was directed at the exposed root of each tooth by marking a single vertical line on a Visual Analogue Scale (VAS) scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm. The score for each participant was calculated by averaging the scores for all study teeth for that participant.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Colgate Regular | Sensodyne Toothpaste | Potassium Oxalate Mouthrinse
Number analyzed (Participants) | 50 | 49 | 50
units on a scale (mm) | 45.41 (2.233) | 32.89 (2.246) | 37.15 (2.227)
Statistical Analysis 1: Comparison: Colgate Regular vs Potassium Oxalate Mouthrinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.010, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean air stimulus VAS score; Mean Difference (Final Values) = -8.26, 95% CI 2-sided [-14.51 to -2.00], Standard Error of Mean 3.163
Statistical Analysis 2: Comparison: Sensodyne Toothpaste vs Potassium Oxalate Mouthrinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.179, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean air stimulus VAS score; Mean Difference (Final Values) = 4.26, 95% CI 2-sided [-1.98 to 10.51], Standard Error of Mean 3.160
Statistical Analysis 3: Comparison: Colgate Regular vs Sensodyne Toothpaste; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean air stimulus VAS score; Mean Difference (Final Values) = -12.52, 95% CI 2-sided [-18.79 to -6.25], Standard Error of Mean 3.172

6. Secondary Outcome: Mean Cold Air Stimulus VAS Score at Week 4
Description: as for outcome 5
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Colgate Regular | Sensodyne Toothpaste | Potassium Oxalate Mouthrinse
Number analyzed (Participants) | 49 | 48 | 50
units on a scale (mm) | 42.03 (2.511) | 24.56 (2.524) | 30.10 (2.479)
Statistical Analysis 1: Comparison: Colgate Regular vs Potassium Oxalate Mouthrinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean air stimulus VAS score; Mean Difference (Final Values) = -11.93, 95% CI 2-sided [-18.93 to -4.93], Standard Error of Mean 3.543
Statistical Analysis 2: Comparison: Sensodyne Toothpaste vs Potassium Oxalate Mouthrinse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.119, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean air stimulus VAS score; Mean Difference (Final Values) = 5.54, 95% CI 2-sided [-1.44 to 12.53], Standard Error of Mean 3.534
Statistical Analysis 3: Comparison: Colgate Regular vs Sensodyne Toothpaste; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Terms included treatment and baseline mean air stimulus VAS score; Mean Difference (Final Values) = -17.47, 95% CI 2-sided [-24.52 to -10.42], Standard Error of Mean 3.566

ADVERSE EVENTS:
Time Frame: Day 28 -2 days/+4 days, +30 days for serious adverse events.
Description: Adverse events were systematically collected at each study visit through Visit 4 (Day 28 -2 days/+4 days). Serious adverse events were reported through 30 days after product use. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Arm/Group | Colgate Regular | Sensodyne Toothpaste | Potassium Oxalate Mouthrinse
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 0/51 | 0/51 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator agreed not to publish the study results without prior sponsor approval.